CLINICAL TRIAL: NCT04407650
Title: Randomised Controlled Trial of Gestational Treatment With Ursodeoxycholic Acid Compared to Metformin to Reduce Effects of Diabetes Mellitus
Brief Title: Ursodeoxycholic Acid vs Metformin in Gestational Diabetes Mellitus
Acronym: GUARD
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 264693
Record Dates: First submitted 2020-05-14; First posted 2020-05-29 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Metformin; Ursodeoxycholic Acid

STUDY DESIGN:
Intervention Model Description: Pilot Phase 4 Randomised Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Active Comparator): Oral 1000 mg BD
  Interventions: Drug: Metformin
- Ursodeoxycholic acid (Experimental): Oral 500 mg BD
  Interventions: Drug: Ursodeoxycholic Acid

INTERVENTIONS:
Drug: Metformin — Patients will be randomized to each intervention using minimisation:
  * BMI category (Overweight/Obese),
  * Previous history of GDM,
  * Disease severity (baseline fasting glucose ≤6.2 or >6.2),
  * Recruitment centre
  Arms: Metformin
Drug: Ursodeoxycholic Acid — Patients will be randomized to each intervention using minimisation:
  * BMI category (Overweight/Obese),
  * Previous history of GDM,
  * Disease severity (baseline fasting glucose ≤6.2 or >6.2),
  * Recruitment centre
  Arms: Ursodeoxycholic acid

SUMMARY:
GUARD is a Clinical Trial that wants to explore the impact of UDCA compared to metformin in the treatment of GDM. The trial wants to recruit 158 women who are overweight or obese who have been diagnosed with GDM, and require pharmacological treatment. Glucose control is our primary measure.

Each year in the UK approximately 35,000 women develop diabetes during pregnancy, a condition called gestational diabetes mellitus (GDM), which increases the risk of adverse outcomes for both mother and child. Metformin, although unlicensed for used in pregnancy, is the most commonly used first line pharmacological treatment. However, there is increasing concern about its widespread use during pregnancy, because of its limited efficacy and because of potential safety concerns. Other common treatments have not been shown to be superior. Therefore, there is an unmet need for additional therapies.

Ursodeoxycholic acid (UDCA) is commonly used in pregnancy for the treatment of intrahepatic cholestasis of pregnancy. It is currently not an established/licensed treatment for GDM. However data from observational studies of women with cholestasis in pregnancy has flagged this to be a potential effective treatment to control blood glucose levels in GDM.

The investigators will ask women to attend three study visits, which will coincide with the time of their antenatal appointments. The trial aims to collect a range of clinical and research blood samples, to measure quality of life and treatment satisfaction through two questionnaires, and will will ask women to wear a continuous glucose monitor for three 10 day periods.

There will be a number of optional assessments that participants will be offered. The primary outcome will be the fasting blood glucose concentration at 36 weeks of gestation.

The investigators intend to carry out this study at 3 sites in the United Kingdom (Guy's and St Thomas, Imperial College and Nottingham), and it has been funded by a J.P Moulton Foundation grant.

DETAILED DESCRIPTION:
GUARD is a two-armed, randomised, controlled, open label multicentre clinical trial with optional observational mechanistic study in a subgroup from each arm, comparing Ursodeoxycholic Acid to Metformin (both oral BD). H0 is no difference in in maternal fasting glucose at 36 weeks. HA is a difference of 6% (0.28mmol/L), consistent with previously reported differences with UDCA treatment for non-alcoholic fatty liver disease (NAFLD). The RCT design was chosen as the generally accepted way of demonstrating clinically important effects of medical treatment, prior to their general acceptance into medical care. The open label is due to the practical difficulty of matching the treatments, due to pill sizes and different dosages.

At present it is known that not all women with GDM respond to oral metformin treatment. Some women cannot tolerate the drug and it is ineffective in others. Many women are reluctant to take insulin as this requires injections and is not without the risk of hypoglycaemia. Therefore there is a need for additional oral treatments to improve glycaemic control. UDCA is a reasonable drug to study as it has good safety data for use in pregnancy (due to studies in women with cholestasis in pregnancy). If previous trials of women with cholestasis is was shown to reduce insulin resistance. It also reduced umbilical cord lipid concentrations. Therefore it is reasonable to compare UDCA to metformin as it may have an equivalent (or better) impact upon glucose control and, if women with GDM have a similar response to those with cholestasis in pregnancy, it could be associated with better outcomes for the baby, e.g. improved umbilical cord blood lipids. As it has not been studied before The investigators do not know if it will be effective, but the existing data suggest it is reasonable to study UDCA. As there is the option of treatment with insulin for women that do not have acceptable glucose control when taking UDCA (as there is for metformin) both drugs are used with an acceptable alternative treatment if they are not sufficiently effective at achieving glycaemic control.

The investigators plan recruitment to last for 18-24 months, and a further 12 months to allow for close out activities.

According to sample size calculations, enrolling 158 participants will provide sufficient statistical power to detect the primary outcome, and allow for a 20% withdrawal rate. An additional 40 participants will be enrolled onto GUARD MEC to serve as controls for this part of the research. Participants will be identified following their OGTT appointment and approached by the diabetes nurse or the study midwife, ideally when they receive dietary and lifestyle education. Interdepartment co-operation will be required.

The Independent Data Monitoring Committee (IDMC) will review outcomes after 25% of the participants have given birth. Data will be monitored by the IDMC at intervals to ensure the interest of participants and validity of data is safeguarded. Most of the outcomes are clinical samples, objective measurements and patient questionnaires. As such researcher bias should have a minimal impact on the reporting. Should this be identified, it will be escalated to the Trial Steering Committee for decision.

An observational sub-study called GUARD MEC will be conducted. 40 GUARD participants, plus other two other control groups (20 women with GDM who do not require pharmacological treatment, and 20 healthy pregnant women), will be invited to participate in the optional study, which will involve eating a specific breakfast in hospital and collecting blood samples at 4 timepoints.

Monitoring of this trial is performed to ensure compliance with Good Clinical Practice, and scientific integrity is managed and oversight retained by the King's Health Partners Clinical Trials Office (KHP-CTO) Quality Team. A study specific monitoring plan has been developed by the KHP-CTO on the basis of a risk assessment. The KHP-CTO will carry out on-site monitoring to undertake source data verification checks and confirm that records are being appropriately maintained by the PI and pharmacy teams.

ELIGIBILITY:
Inclusion Criteria:

1. Women between 16 and 45 years of age with GDM diagnosed at 26+0 to 30+6 weeks' gestation in accordance with the NICE guidelines (one or more glucose concentrations of ≥5.6 mmol/l fasting or ≥7.8 mmol/l 2 hours after a standard 75g OGTT, and requiring pharmacological treatment).
2. Overweight or obese (Booking BMI ≥25 kg/m2)
3. Planned antenatal, intrapartum and postpartum care at the participating centre (i.e. not planning to move before delivery).

Exclusion Criteria:

1. Unwilling/unable to give written informed consent and comply with the requirements of the study protocol
2. Multiple pregnancies (twins, triplets etc) in current pregnancy
3. Congenital anomaly on ultrasound requiring fetal medicine input
4. Previous diagnosis of diabetes outside pregnancy
5. HbA1c at booking >48 mmol/mol or ≥6.5% during current pregnancy (if available)
6. Significant pre-pregnancy comorbidities that increase risk in pregnancy, for example renal failure, severe liver disease, transplantation, cardiac failure, psychiatric conditions requiring in-patient admission (within previous year) in the opinion of the responsible clinician or the CI.
7. Significant co-morbidity in the current pregnancy, nephropathy (estimated GFR <60ml/min), other physical or psychological conditions likely to interfere with the conduct of the study and/or interpretation of the trial results in the opinion of the responsible clinician or the CI.
8. Not fluent in English and absence of interpreter or translation services (ie telephone translation services)
9. Participating in another intervention study where the results could influence GDM-related endpoints, in the opinion of the responsible clinician or the CI, or participation in a CTIMP during current pregnancy.
10. Known allergy/hypersensitivity/intolerance to the active substance or excipients, or patients taking any medications which are contraindicated as per IMP SmPC

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Only pregnant people allowed study entry, irrespective of gender indentity
Enrollment: 64 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Glycaemic control | Gestational week 36
  Maternal fasting glucose concentration in blood sample

SECONDARY OUTCOMES:
Acceptability | Gestational week 36
  To assess the acceptability of UDCA compared to metformin using the Diabetes Treatment Satisfaction Questionnaire GB-DTSQs_Jul94 with scales ranging from 6 (increased satisfaction/acceptability) - 0 (dissatisfaction)
Biomedical outcomes: continuous glucose monitoring | Baseline (week 28), Follow up 1 (week 32), Follow up 2 (week 36)
  Glucose metabolism control measured by continuous glucose monitors to establish whether continuous glucose monitoring gives more informative overall assessment of maternal glycaemic control
Biomedical outcomes: 1,5-anhydroglucitol | Baseline (week 28), Follow up 1 (week 32), Follow up 2 (week 36)
  Glucose metabolism control measured by serum concentrations of 1,5-anhydroglucitol
Biomedical outcomes: glucose control by HbA1c | Baseline (week 28), Follow up 2 (week 36)
  Glucose metabolism control measured by HbA1c concentration
Biomedical outcomes: lipids | Follow up 2 (week 36)
  Lipid metabolism assessed by blood triglyceride, total cholesterol, calculated LDL-cholesterol, HDL-cholesterol and free fatty acid concentrations, all in mmol/L
Biomedical analyses: bilirubin | Follow up 2 (week 36)
  Maternal liver function tests: bilirubin
Biomedical analyses: ALT | Follow up 2 (week 36)
  Maternal liver function tests: ALT
Biomedical analyses: bile acids | Follow up 2 (week 36)
  Maternal liver function tests: bile acids
Biomedical analyses: CRP | Follow up 2 (week 36)
  Maternal liver function tests: C reactive protein
Clinical maternal outcomes: insulin | From enrolment to birth
  Proportion of women requiring insulin treatment (time until treatment and dose)
Clinical maternal outcomes: weight | Follow up 2 (week 36) compared to first trimester
  Maternal weight change
Maternal vascular responses (I) | Follow up 1 (week 32), Follow up 2 (week 36)
  maternal pulse wave velocity (PWV)
Maternal vascular responses (II) | Follow up 1 (week 32), Follow up 2 (week 36)
  systolic and diastolic blood pressure
Maternal vascular responses (III) | Follow up 1 (week 32), Follow up 2 (week 36)
  central arterial pressure (cP)
Maternal vascular responses (IV) | Follow up 1 (week 32), Follow up 2 (week 36)
  Augmentation index (AIx)
Blood loss | Delivery
  Estimated blood loss during birth
Neonatal outcomes: mode of birth | Delivery
  Amongts all participants, caesarean section (elective & emergency), assisted vaginal birth and spontaneous vaginal delivery numbers will be measured
Neonatal outcomes: gestational age | Delivery
  Gestational age at birth
Neonatal outcomes: apgar scores | Delivery
  Apgar scores at 5 minutes post birth
Neonatal outcomes: shoulder dystocia | Delivery
  Occurrence of shoulder dystocia
Neonatal outcomes: weight | Delivery
  Infant birth weight will be collected to analyse the percentage proportion of babies born large for gestational age and proportion of babies born small for gestational age
Neonatal outcomes: morbidity | Delivery
  Treatment for neonatal hypoglycaemia, neonatal jaundice, respiratory distress or birth trauma
Neonatal outcomes: rate of special care unit admission. | 28 days post delivery
  Neonatal intensive care and special care unit admission (duration of hospital stay)
Stillbirth and neonatal death | Delivery
  Occurrence of stillbirth and neonatal death
Biomedical neonatal outcomes | Delivery
  Cord blood C-peptide, triglyceride, total cholesterol, calculated LDL-cholesterol, HDL-cholesterol and free fatty acid concentrations all in mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Ovadia, CI, Principal Investigator — King's College London
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lovell H, Mitchell A, Ovadia C, Pitrelli N, Briley A, Singh C, Marschall HU, Cruickshank K, Murphy H, Seed P, Williamson C. A multi-centered trial investigating gestational treatment with ursodeoxycholic acid compared to metformin to reduce effects of diabetes mellitus (GUARD): a randomized controlled trial protocol. Trials. 2022 Jul 19;23(1):571. doi: 10.1186/s13063-022-06462-y. PMID 35854327

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/50/NCT04407650/Prot_SAP_000.pdf